CLINICAL TRIAL: NCT05209308
Title: A Phase 2 Single-Arm, Open-Label Study to Assess the Safety and Efficacy of Rituximab Plus Venetoclax in Combination With Zandelisib in Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia - The CORAL Study
Brief Title: Rituximab Plus Venetoclax in Combination With Zandelisib in Subjects With CLL
Acronym: CORAL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Discontinuation of zandelisib development
Sponsor: MEI Pharma, Inc. (Industry)
Collaborators: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ME-401-008
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: CLL
Keywords: Leukemia
MeSH Terms: conditions — Leukemia | interventions — ME-401; Rituximab; venetoclax

STUDY DESIGN:
Intervention Model Description: This open label study is composed of 2 cohorts:
  A safety run-in Cohort A followed by Cohort B.
  Both cohorts will follow the same dosing schedule and subjects will receive Zandelisib, however in Cohort A, VEN will be administered at a different dose then Cohort B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Ven "low dose" + Rituximab + Zandelisib
  Interventions: Drug: Zandelisib; Drug: Rituximab; Drug: Venetoclax
- Cohort B (Experimental): Ven "standard dose" + Rituximab + Zandelisib
  Interventions: Drug: Zandelisib; Drug: Rituximab; Drug: Venetoclax

INTERVENTIONS:
Drug: Zandelisib — Zandelisib taken orally for 7 days of each 28 day cycle
  Other Names: ME-401
Drug: Rituximab — Rituximab IV for 6 cycles
  Other Names: Rituxan; MabThera
Drug: Venetoclax — Orally - Ramp up weeks 1-5
  Other Names: Venclexta

SUMMARY:
A Phase 2 study of Zandelisib with Venetoclax (VEN) and Rituximab (R) in subjects with Relapsed/Refractory CLL.

DETAILED DESCRIPTION:
This is an open label Phase 2 clinical study of Zandelisib with Venetoclax (VEN) and Rituximab (R) in subjects with R/R CLL.

VEN and R will be administered per standard of care.

Subjects must have histologically confirmed relapsed/refractory CLL and received ≥1 lines of prior therapy

A total 42 subjects will be enrolled and treated with zandelisib in combination with VEN + R.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥18 years
* Histologically confirmed relapsed/refractory CLL who received ≥1 lines of prior therapy
* At least one bi-dimensionally measurable nodal lesion >1.5 cm
* Adequate renal, hepatic function
* Adequate hematologic parameters at screening

Exclusion Criteria:

* Subjects who relapsed or progressed on BCL-2 inhibitor
* Relapsed within 2 years of discontinuation of prior PI3K inhibitor (PI3Ki) therapy or disease progression on PI3Ki therapy
* History or currently active HBV, HCV; any uncontrolled active infection, HIV infection; HIV-related lymphoma
* History of Richter's transformation or prolymphocytic leukemia
* Known allergies to both xanthine oxidase inhibitors and rasburicase, or any excipients of the drug products
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
To determine the uMRD rate in PB and BM by flow cytometry | 2 year
  measured by 8-color flow cytometry with a quantitative lower limit of detection of at least 10-4 (1 in 10,000 cells).

SECONDARY OUTCOMES:
ORR | 2 years
  The ORR will be measured by the proportion of subjects having achieved a CR/CRi (CR with incomplete recovery in BM) or partial response (PR) according to the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) guidelines (2018)
Progression Free Survival | 5 years
  PFS will be measured as the time from first dose date until progression according the iwCLL criteria or death from any cause.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Stony Brook University, Stony Brook, New York
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Medical Oncology Associates, PS (dba Summit Cancer Centers), Spokane, Washington